CLINICAL TRIAL: NCT06199232
Title: Targeted Treatment Based on ctDNA Genotyping Combined With Tislelizumab and HAIC as Salvage Treatment for Advanced Colorectal Cancer Liver Metastasis Failed From Standard Systemic Treatment (SALVLIV Trial)
Brief Title: Targeted Treatment Plus Tislelizumab and HAIC for Advanced CRCLM Failed From Standard Systemic Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SALVLIVE
Record Dates: First submitted 2023-12-24; First posted 2024-01-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Liver Metastasis Colon Cancer; ctDNA Genotype; MSS; Failed From Standard Treatment
Keywords: hepatic arterial infusion chemotherapy; targeted therapy; tislelizumab; ctDNA genotype; MSS CRCLM

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): HAIC combined with targeted therapy and PD-1 inhibitor
  Interventions: Drug: HAIC+targeted therapy+PD-1 inhibitor

INTERVENTIONS:
Drug: HAIC+targeted therapy+PD-1 inhibitor — HAIC regimen: doublet or triplet regimen based on the response and adverse events occurred in the previous standard treatment (depended on the decision of researchers)-oxaliplatin (85 mg/m2, split into d1 and d2, 0-2h,) and 5-fluorouracial (2g/m2, split into d1 and d2, 2-24h)/ oxaliplatin (65 mg/m2, 0-2h, d1), irinotecan (100 mg/m2, 0-2h, d2), and 5-fluorouracial (2g/m2, split in d1 and d2, 2-24h), repeated every 4 weeks; drug-eluting TACE will be performed at 3rd-4th cycles if the lesions in liver is abundant with blood supply.
  Tislelizumab (a PD-1 inhibitor): 200 mg, intravenous drip for 30-60 minutes before 24h of HAIC, q4w.
  Cetuximab (Group A, KRAS/NRAK/BRAF/EGFR wide type and interrupt cetuximab more than 3 months): 500 mg/m2, intravenous drip before HAIC, q4w.
  Fruquintinib (Group B, KRAS/NRAS/BRAF/EGFR mutation type and wide type but treated with cetuximab in last 3 months): 3 mg/d, d3-23, then suspend for 1w.
  Other Names: HAIC+Fruquintinib/Cetuximab+Tislelizumab

SUMMARY:
Hepatic arterial infuison chemothearpy (HAIC), targeted therapy, and programmed death-1 (PD-1) inhibitors have been demonstrated to be effective for colorectal cancer liver metastasis (CRCLM). Thus, the investigators will conduct a prospective trial to explore the efficacy and safety of targeted treatment based on ctDNA genotyping combined with tislelizumab and HAIC as salvage treatment for advanced CRCLM failed from standard systemic treatment, aiming to provide individualized optimized regimen for microsatellite stable (MSS) CRCLM in salvage treatment.

DETAILED DESCRIPTION:
Although surgery has been demonstrated to improve the prognosis of patients with colorectal cancer liver metastasis (CRCLM), only 20% of patients with CRCLM is candidate for surger. Irinotecan-/oxaliplatin-based doublet/triplet chemotherapy regimen combined with targeted therapy (anti vascular endothelial growth factor [VEFG] or anti epidermal growth factor receptor [EGFR]) based on the genotype are recommended as standard first- and second-line treatment for unresectabel metastatic colorectal cancer (mCRC) by NCCN guideline. RAS and BRAF are the important signal members in the EGFR signal pathway, and the mutation of them could induce the persistent activation of the downstream of the MAPK pathway, leading to the differentiation, proliferation, and growth change of the tumor cell. The status of RAS and BRAF V600E mutation will affect the efficacy of anti-EGFR therapy, but not anti-VEGF therapy.

Regorafenib, fruquintinb, and TAS-102 have been recommended as third-line treatment for mCRC, while the survivl benefits from these agents are limited, with the median progression-free survival (PFS) and median OS of 1.9-3.7 months and 6.4-9.3 months, respectively.

The efficacy and safety of hepatic arterial infusion chemotherapy (HAIC) for CRCLM have been demonstrated by multiple trials and recommended by many guidelines worldwide. Fruquintinib, a small molecular tyrosine kinase inhibitor targeting at VEGF 1-3, has been demonstrated to change the tumor microenvironment and enhance the anti-tumor effect of programmed death-1 (PD-1) inhibitor in microsatellite stable (MSS) CRC. Anti-EGFR rechallenge (cetuximab rechallenge) was effective in patients with CRC who interrupted the anti-EGFR therapy while responsed to anti-EGFR therapy in the first-line treatment. In 2021, a phase II trial, which explore the efficacy and safety of cetuximab rechallenge combined with Avelumab for pretreated RAS wide type (WT) mCRC. Our retrospective study (unpublished) showed HAIC combined with fruquintinib and tislelizumab presented greater efficacy for MSS CRCLM.

Thus, the investigators will conduct a prospective trial to explore the efficacy and safety of targeted treatment based on ctDNA genotyping combined with tislelizumab and HAIC as salvage treatment for advanced CRCLM failed from standard systemic treatment, aiming to provide individualized optimized regimen for MSS CRCLM in salvage treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old.
2. Colorectal cancer confirmed by histopatology.
3. The metastasis is mainly located in liver.
4. Unresectable liver metastasis is confirmed by CT/MRI scan and multidisciplinary.
5. Failed from standard first- and second-line systemic treatment.
6. At least one measurable lesion according to modified Response Evaluation Criteria in Solid Tumors guidelines (mRECIST).
7. Eastern Cooperative Oncology Group (ECOG) performance status <2.
8. Child-Pugh A or B (≤ 7).
9. Expectant survival time ≥ 3 months.
10. Adequate organ function as follows:

    1. Hemoglobin ≥ 90 g/L;
    2. Absolute neutrophil count ≥ 1.5×10^9/L;
    3. Blood platelet count ≥ 775×10^9/L;
    4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 5 times of upper limit of normal (ULN);
    5. Total bilirubin ≤ 2 times of ULN;
    6. Serum creatinine ≤ 1.5 times of ULN;
    7. Albumin ≥ 30 g/L.
11. Patients sign informed consent.

Exclusion Criteria:

1. Extensive extrahepatic metastasis (>25% of tumor burden in liver).
2. HER2 (3+) or HER2 amplification.
3. MSI-H or dMMR.
4. Allergic to contrast media.
5. Pregnant or lactational.
6. Allergic to oxaliplatin or cetuximab.
7. Coinstantaneous a lot of malignant hydrothorax or ascites.
8. History of organ transplantation (including bone marrow auto-transplantation and peripheral stem cell transplantation).
9. Coinstantaneous infection and need anti-infection therapy.
10. Coinstantaneous peripheral nervous system disorder.
11. History of obvious mental disorder and central nervous system disorder.
12. Concomitant malignancy within 5 years, except for non-melanoma skin cancer and carcinoma in situ of cervix.
13. Without legal capacity.
14. Impact the study because of medical or ethical reasons.
15. Clinically severe gastrointestinal bleeding within 6 months of the start of treatment or any life-threatening bleeding events within 3 months of the start of treatment.
16. Uncorrectable coagulation disorder.
17. Obvious abnormal in ECG or obvious clinical symptoms of heart disease, like congestive heart failure, coronary heart disease with obvious clinical symptoms, unmanageable arrhythmia and hypertension.
18. History of myocardial infarction within 12 months, or Grade III/IV of heart function.
19. Severe liver disease (like cirrhosis), renal disease, respiratory disease, unmanageable diabetes or other kinds of systematic disease.
20. Any other subjects that the investigator considers ineligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2027-05-23 (Estimated)

PRIMARY OUTCOMES:
PFS rate at 6 months | From the date of treatment begining to the date of 6 months after the treatment begining.
  Proportion of patients with 6- month progression-free survival after treatment begining in all patients.

SECONDARY OUTCOMES:
PFS | From date of treatment beginning until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The time from treatment initiation to the first documented disease progression or death due to any cause, whichever occurs firstly
OS | From date of treatment beginning until the date of death from any cause, assessed up to 100 months
  The time from treatment initiation to death due to any cause
intrahepatic PFS | From date of treatment beginning until the date of first documented progression in liver or date of death from any cause, whichever came first, assessed up to 100 months
  The time from treatment initiation to the first documented disease progression in liver or death due to any cause, whichever occurs firstly
ORR | Evaluation of tumor burden based on mRECIST criteria through study completion, an average of once per 3 months.
  The proportion of participants in the analysis population who have complete response (CR) or partial response (PR) determined by investigators using mRECIST criteria at any time during the study.
DCR | Evaluation of tumor burden based on mRECIST criteria through study completion, an average of once per 3 months.
  The proportion of participants in the analysis population who have complete response (CR), partial response (PR), or stable disease (SD) determined by investigators using mRECIST criteria at any time during the study.
Number of patients with treatment-related adverse events | Through study completion, an average of once per 1 month.
  Number of patients with AE, treatment-related AE (TRAE), serious adverse event (SAE) assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Wang, M.D., Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peking Univerisity Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanas GP, Taylor A, Primrose JN, Langeberg WJ, Kelsh MA, Mowat FS, Alexander DD, Choti MA, Poston G. Survival after liver resection in metastatic colorectal cancer: review and meta-analysis of prognostic factors. Clin Epidemiol. 2012;4:283-301. doi: 10.2147/CLEP.S34285. Epub 2012 Nov 7. PMID 23152705
- [Background] Hackl C, Neumann P, Gerken M, Loss M, Klinkhammer-Schalke M, Schlitt HJ. Treatment of colorectal liver metastases in Germany: a ten-year population-based analysis of 5772 cases of primary colorectal adenocarcinoma. BMC Cancer. 2014 Nov 4;14:810. doi: 10.1186/1471-2407-14-810. PMID 25369977
- [Background] Cho M, Gong J, Fakih M. The state of regional therapy in the management of metastatic colorectal cancer to the liver. Expert Rev Anticancer Ther. 2016;16(2):229-45. doi: 10.1586/14737140.2016.1129277. Epub 2016 Jan 13. PMID 26652741
- [Background] Wang Y, Wei B, Gao J, Cai X, Xu L, Zhong H, Wang B, Sun Y, Guo W, Xu Q, Gu Y. Combination of Fruquintinib and Anti-PD-1 for the Treatment of Colorectal Cancer. J Immunol. 2020 Nov 15;205(10):2905-2915. doi: 10.4049/jimmunol.2000463. Epub 2020 Oct 7. PMID 33028620
- [Background] Li Q, Cheng X, Zhou C, Tang Y, Li F, Zhang B, Huang T, Wang J, Tu S. Fruquintinib Enhances the Antitumor Immune Responses of Anti-Programmed Death Receptor-1 in Colorectal Cancer. Front Oncol. 2022 Mar 17;12:841977. doi: 10.3389/fonc.2022.841977. eCollection 2022. PMID 35371995
- [Result] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Result] Li J, Qin S, Xu R, Yau TC, Ma B, Pan H, Xu J, Bai Y, Chi Y, Wang L, Yeh KH, Bi F, Cheng Y, Le AT, Lin JK, Liu T, Ma D, Kappeler C, Kalmus J, Kim TW; CONCUR Investigators. Regorafenib plus best supportive care versus placebo plus best supportive care in Asian patients with previously treated metastatic colorectal cancer (CONCUR): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2015 Jun;16(6):619-29. doi: 10.1016/S1470-2045(15)70156-7. Epub 2015 May 13. PMID 25981818
- [Result] Li J, Qin S, Xu RH, Shen L, Xu J, Bai Y, Yang L, Deng Y, Chen ZD, Zhong H, Pan H, Guo W, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Chen D, Li W, Sun S, Yu Z, Cao P, Chen H, Wang J, Wang S, Wang H, Fan S, Hua Y, Su W. Effect of Fruquintinib vs Placebo on Overall Survival in Patients With Previously Treated Metastatic Colorectal Cancer: The FRESCO Randomized Clinical Trial. JAMA. 2018 Jun 26;319(24):2486-2496. doi: 10.1001/jama.2018.7855. PMID 29946728
- [Result] Mayer RJ, Van Cutsem E, Falcone A, Yoshino T, Garcia-Carbonero R, Mizunuma N, Yamazaki K, Shimada Y, Tabernero J, Komatsu Y, Sobrero A, Boucher E, Peeters M, Tran B, Lenz HJ, Zaniboni A, Hochster H, Cleary JM, Prenen H, Benedetti F, Mizuguchi H, Makris L, Ito M, Ohtsu A; RECOURSE Study Group. Randomized trial of TAS-102 for refractory metastatic colorectal cancer. N Engl J Med. 2015 May 14;372(20):1909-19. doi: 10.1056/NEJMoa1414325. PMID 25970050